CLINICAL TRIAL: NCT01277159
Title: Duration of Analgesia After Popliteal Fossa Nerve Blockade: Effects of Dexamethasone and Buprenorphine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2012-042
Record Dates: First submitted 2011-01-13; First posted 2011-01-14 (Estimated); Results first posted 2017-08-31 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Patients Undergoing Ankle Surgery
Keywords: Analgesia; Duration; Popliteal Fossa Nerve Block; Dexamethasone; Buprenorphine; Additives; Ankle surgery
MeSH Terms: conditions — Agnosia | interventions — Dexamethasone; Sodium Chloride; Buprenorphine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Control Nerve Block. IV Dexamethasone (4 mg). (Experimental): Control Nerve Block. IV Dexamethasone (4 mg).
  Interventions: Drug: A. Control Nerve Block. IV Dexamethasone (4 mg).
- Nerve Block with Dexamethasone (4 mg). IV saline. (Experimental): B. Nerve Block with Dexamethasone (4 mg). IV saline.
  Interventions: Drug: B. Nerve Block with Dexamethasone (4 mg). IV saline.
- Control Nerve Block. IV Dexamethasone (4 mg). IV Buprenorp (Experimental): Control Nerve Block. IV Dexamethasone (4 mg). IV Buprenorphine (0.3 mg)
  Interventions: Drug: C. Control Nerve Block. IV Dexamethasone (4 mg). IV Buprenorphine (0.3 mg)
- Nerve Block with Buprenorphine (0.3 mg). IV Dexamethasone ( (Experimental): Nerve Block with Buprenorphine (0.3 mg). IV Dexamethasone (4 mg).
  Interventions: Drug: D. Nerve Block with Buprenorphine (0.3 mg). IV Dexamethasone (4 mg).
- Nerve Block with Dexamethasone (4 mg) / block Buprenorphine (Experimental): Nerve Block with Dexamethasone (4 mg) / block Buprenorphine (0.3 mg). IV saline.
  Interventions: Drug: E. Nerve Block with Dexamethasone (4 mg) / block Buprenorphine (0.3 mg).

INTERVENTIONS:
Drug: A. Control Nerve Block. IV Dexamethasone (4 mg). — A. Control Nerve Block. IV Dexamethasone (4 mg).
  Arms: Control Nerve Block. IV Dexamethasone (4 mg).
Drug: B. Nerve Block with Dexamethasone (4 mg). IV saline. — B. Nerve Block with Dexamethasone (4 mg). IV saline.
  Arms: Nerve Block with Dexamethasone (4 mg). IV saline.
Drug: C. Control Nerve Block. IV Dexamethasone (4 mg). IV Buprenorphine (0.3 mg) — C. Control Nerve Block. IV Dexamethasone (4 mg). IV Buprenorphine (0.3 mg)
  Arms: Control Nerve Block. IV Dexamethasone (4 mg). IV Buprenorp
Drug: D. Nerve Block with Buprenorphine (0.3 mg). IV Dexamethasone (4 mg). — D. Nerve Block with Buprenorphine (0.3 mg). IV Dexamethasone (4 mg).
  Arms: Nerve Block with Buprenorphine (0.3 mg). IV Dexamethasone (
Drug: E. Nerve Block with Dexamethasone (4 mg) / block Buprenorphine (0.3 mg). — E. Nerve Block with Dexamethasone (4 mg) / block Buprenorphine (0.3 mg). IV saline.
  Arms: Nerve Block with Dexamethasone (4 mg) / block Buprenorphine

SUMMARY:
Patients scheduled to go home after ankle surgery at HSS typically receive a sciatic nerve block in the popliteal fossa and oral analgesic tablets (such as Percocet). Popliteal fossa nerve blockade has reduced pain for these patients (YaDeau et al, Anesth Analg 2008;106:1916-20), but unfortunately the patients still often experience moderate to severe pain after the block wears off. The investigators wish to study two additives that may prolong the period of analgesia provided by the nerve block. The additives will be studied in the context of a standardized postoperative multimodal analgesic pathway.

Primary outcome:

Does adding dexamethasone and / or buprenorphine prolong the analgesia provided by a popliteal fossa nerve block?

ELIGIBILITY:
Inclusion Criteria:

1. Patients of Dr Levine or Dr Roberts.
2. Scheduled for discharge from HSS after foot or ankle surgery.
3. A single-injection popliteal fossa nerve block is judged appropriate.
4. Surgery confined to foot and ankle (no iliac crest bone graft planned - iliac aspirate is not an exclusion criterion).
5. Patients aged 18-75 years.

Exclusion Criteria:

* Surgery that will cause pain at sites outside the distal lower extremity (e.g. iliac crest bone graft).
* Bilateral surgery
* Chronic pain (defined as regular use of opioid analgesics for > 3 months).
* Chronic use of steroids (defined as regular use of steroids for > 3 months).
* Contraindication to performance of the popliteal fossa nerve block with 30 cc 0.25% bupivacaine with clonidine (e.g. alleged bupivacaine sensitivity, low body weight, clonidine allergy, etc.).
* Contraindications to dexamethasone or buprenorphine (e.g. allergy, Insulin Dependent Diabetes Mellitus, etc.)
* Inability of the patient to describe postoperative pain (e.g. psychiatric disorder, dementia).
* Non-English speaking patients (the questionnaire is in English, and translations would have to be separately validated)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2010-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Urban, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Nerve Block With Dexamethasone (4 mg) / Block Buprenorphine: Nerve Block with Dexamethasone (4 mg) / block Buprenorphine (0.3 mg). IV saline.
  E. Nerve Block with Dexamethasone (4 mg) / block Buprenorphine (0.3 mg).: E. Nerve Block with Dexamethasone (4 mg) / block Buprenorphine (0.3 mg).
  IV saline.
Period: Overall Study
Arm/Group | Control Nerve Block. IV Dexamethasone (4 mg). | Nerve Block With Dexamethasone (4 mg). IV Saline. | Control Nerve Block. IV Dexamethasone (4 mg). IV Buprenorp | Nerve Block With Buprenorphine (0.3 mg). IV Dexamethasone ( | Nerve Block With Dexamethasone (4 mg) / Block Buprenorphine
Started | 21 | 22 | 22 | 22 | 21
Completed | 17 | 21 | 19 | 19 | 16
Not Completed | 4 | 1 | 3 | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Nerve Block. IV Dexamethasone (4 mg). | Nerve Block With Dexamethasone (4 mg). IV Saline. | Control Nerve Block. IV Dexamethasone (4 mg). IV Buprenorp | Nerve Block With Buprenorphine (0.3 mg). IV Dexamethasone ( | Nerve Block With Dexamethasone (4 mg) / Block Buprenorphine | Total
Number analyzed (Participants) | 17 | 21 | 19 | 19 | 16 | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.29 (6.8) | 47.81 (9.5) | 46.26 (7.5) | 47.95 (8.6) | 52.19 (7.2) | 49.1 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 13 | 10 | 14 | 13 | 61
  Male | 6 | 8 | 9 | 5 | 3 | 31
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Time it Takes for Nerve Block to Wear Off
Description: Does adding dexamethasone and / or buprenorphine prolong the analgesia provided by a popliteal fossa nerve block?
Time Frame: up to 72 hours
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Control Nerve Block. IV Dexamethasone (4 mg). | Nerve Block With Dexamethasone (4 mg). IV Saline. | Control Nerve Block. IV Dexamethasone (4 mg). IV Buprenorp | Nerve Block With Buprenorphine (0.3 mg). IV Dexamethasone ( | Nerve Block With Dexamethasone (4 mg) / Block Buprenorphine
Number analyzed (Participants) | 17 | 21 | 19 | 19 | 16
hours | 30.4 (5.1) | 45.1 (5.2) | 32.2 (6.1) | 45.6 (5.6) | 45.6 (5.8)

ADVERSE EVENTS:
Arm/Group | Control Nerve Block. IV Dexamethasone (4 mg). | Nerve Block With Dexamethasone (4 mg). IV Saline. | Control Nerve Block. IV Dexamethasone (4 mg). IV Buprenorp | Nerve Block With Buprenorphine (0.3 mg). IV Dexamethasone ( | Nerve Block With Dexamethasone (4 mg) / Block Buprenorphine
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/21 | 0/19 | 0/19 | 0/16
Other Adverse Events (participants affected / at risk) | 0/17 | 0/21 | 0/19 | 0/19 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes